CLINICAL TRIAL: NCT05562492
Title: An Open-label, Multi-centre, Randomised, Two Arm Single Period Parallel Study to Assess the Efficacy, Safety and Utility of Hybrid Closed-loop Glucose Control Compared to Standard Insulin Therapy Combined With Continuous Glucose Monitoring in Young People (≥16 Years) and Adults With Cystic Fibrosis Related Diabetes (CL4P-CF Study)
Brief Title: Closed-loop for People Living With Cystic Fibrosis Related Diabetes
Acronym: CL4P-CF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: University of Oxford (Other); University of Edinburgh (Other)
Responsible Party: Principal Investigator, Dr Charlotte Boughton, Clinical Lecturer, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL4P-CF
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis-related Diabetes
Keywords: closed-loop
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: An open-label, multicentre, randomised, two-arm single-period parallel design study contrasting closed-loop insulin therapy and standard insulin therapy with CGM in young people (≥16 years) and adults with CF related diabetes over 26 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed-loop insulin delivery (CamAPS FX) (Experimental): The automated closed loop system (CamAPS FX) will consist of:
  YpsoPump insulin pump (Ypsomed, Burgdorf, Switzerland) Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA) A smartphone hosting CamAPS FX app with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump and glucose sensor Cloud upload system to review CGM/insulin data.
  Participants will use the closed-loop system for the next 26 weeks at home
  Interventions: Device: CamAPS FX
- Conventional insulin therapy with CGM (Active Comparator): Usual insulin therapy (injections or pump) and study CGM for 26 weeks at home.
  Interventions: Other: Standard insulin therapy with CGM

INTERVENTIONS:
Device: CamAPS FX — The automated closed loop system (CamAPS FX) will consist of:
  YpsoPump insulin pump (Ypsomed, Burgdorf, Switzerland) Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA) An Android smartphone hosting CamAPS FX app with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump and glucose sensor Cloud upload system to review CGM/insulin data.
  Arms: Closed-loop insulin delivery (CamAPS FX)
Other: Standard insulin therapy with CGM — Usual insulin therapy and study CGM.
  Arms: Conventional insulin therapy with CGM

SUMMARY:
The main objective of this study is to determine whether closed-loop glucose control is superior to standard insulin therapy with continuous glucose monitoring (CGM) in young people (≥16 years) and adults with cystic fibrosis (CF) related diabetes.

This is an open-label, multicentre, randomised, single-period, two-arm parallel design study, involving a run-in period followed by a 26 week intervention period during which glucose levels will be controlled either by a hybrid closed-loop system or by participants usual insulin therapy with continuous glucose monitoring. A total of up to 128 young people and adults (aiming for 114 completed participants) with CF related diabetes using insulin will be recruited through outpatient CF and diabetes clinics and other established methods at participating centres. Participants who drop out of the study within the first 4 weeks of the intervention period will be replaced.

Participants will receive appropriate training in the safe use of the CGM and closed-loop devices. Participants will have access to the study team during the intervention phase with 24/7 telephone support.

The primary outcome is time spent in target range between 3.9 and 10.0 mmol/L as recorded by CGM over the 26 week period. Other key endpoints include time above target glucose range (>10mmol/L), mean glucose, and HbA1c. Secondary outcomes include time spent with glucose levels below target as recorded by CGM, and other CGM-based metrics in addition to percent of predicted FEV1, body mass index, fasting C-peptide levels, insulin requirements and number of pulmonary exacerbations and hospitalisations. Safety evaluation comprises severe hypoglycaemic episodes, and other adverse and serious adverse events.

Psychosocial outcomes include CGM & closed-loop usage, health-related quality of life questionnaires, burden of diabetes management assessment and semi-structured interviews after participants have had at least three months experience of using the technology. Data will be collected for future health economic analysis.

DETAILED DESCRIPTION:
Purpose of clinical trial:

To determine if closed-loop can improve glucose control and health-related quality of life compared to standard insulin therapy with CGM in young people (≥16 years) and adults with Cystic Fibrosis related diabetes.

Study objectives:

The study objective is to compare closed-loop glucose control with standard insulin therapy with CGM in young people and adults with CF related diabetes in terms of:

1. EFFICACY:

   * GLYCAEMIC CONTROL: The objective is to assess the efficacy of closed-loop in maintaining CGM glucose levels within the target range from 3.9 to 10.0 mmol/l, as compared to standard insulin therapy combined with CGM (primary endpoint) and other measures of glucose control.
   * LUNG FUNCTION: frequency of pulmonary exacerbations, hospitalisations and forced expiratory volume in 1 second (FEV1).
   * METABOLIC: body mass index (BMI) and endogenous insulin secretion (C-peptide).
   * HEALTH-RELATED QUALITY OF LIFE: CF-specific and generic measures and interviews to assess psychosocial aspects and responses of participants to the technology.
2. SAFETY:

   The objective is to evaluate the safety of closed-loop glucose control in terms of episodes of severe hypoglycaemia and other adverse events and adverse device effects.
3. ACCEPTABILITY:

   The objective is to determine the duration of use of CGM and closed-loop, and usability and acceptance of the closed-loop system.
4. HEALTH ECONOMIC:

The objective is to determine the clinical and cost effectiveness of closed-loop in the patient population compared with current standard care from the perspective of the NHS and social services.

Participating clinical centres:

Addenbrooke's Hospital, Cambridge University Hospital NHS Foundation Trust, UK Royal Papworth Hospital, Cambridge, UK Royal Brompton Hospital, London, UK Wythenshawe Hospital, Manchester University NHS Foundation Trust, UK Kings College Hospital, London, UK Birmingham Heartlands Hospital, University Hospitals Birmingham NHS Foundation Trust, UK Churchill Hospital, Oxford University Hospital NHS Foundation Trust, UK

Sample Size:

114 young people (≥16 years) and adults completing the study. Up to 128 participants will be recruited to allow for dropouts.

Maximum duration of study for a subject: 28 weeks (7 months)

Recruitment:

Participants will be recruited through outpatient CF or diabetes clinics or other established methods at participating centres.

Consent:

Participants will be asked to provide written informed consent.

Baseline Assessment:

Eligible participants will undergo a baseline evaluation involving taking a medical history including demographics, CF characteristics, genotype and current therapies, height/weight, spirometry (FEV1) and blood samples including HbA1c, C-peptide and glucose. Urine pregnancy test will be done in females of child-bearing age. Validated questionnaires will be completed and a masked glucose sensor applied.

Run-in Period:

During the 2-3 week run-in period, participants will use their own insulin therapy and wear a masked CGM system. At the end of the run-in period, for compliance, at least 10 days of CGM data needs to be recorded. CGM data during the run-in period will be used to assess baseline glucose control before the start of the intervention phase. Only those with time in target glucose range <80% during this period will proceed to randomisation.

Randomisation:

Eligible participants will be randomised in a 1:1 ratio using central randomisation software to the use of closed-loop or to standard therapy with CGM for 26 weeks. Randomisation will be stratified by site, age and baseline time in target glucose range.

Automated closed loop insulin delivery (intervention arm):

Training on the use of closed-loop will be provided by the research team during a 1 to 2 hour session in an outpatient setting (clinical research facility) or may be done remotely. Competency on the use of study insulin pump, study CGM and closed-loop system will be evaluated using a competency assessment tool developed by the research team. Further training may be delivered as required. Participants will be advised to use the closed-loop system for the next 26 weeks at home.

Conventional insulin therapy with CGM (control arm):

Participants will use their own insulin therapy (injections or pump) and study CGM. Training on the use of real-time CGM and how to interpret real-time will be provided. Participants will use standard insulin therapy and real-time CGM for the next 26 weeks at home.

3 month study visit: The following measurements will be taken: weight, spirometry (FEV1) and blood samples including HbA1c, C-peptide and glucose. Data from the closed-loop system and CGM system will be reviewed. Validated questionnaires will be completed.

End of study assessments:

The following measurements will be taken: weight, spirometry (FEV1) and blood samples including HbA1c, C-peptide and glucose. Data from the closed-loop system and CGM system will be reviewed. Validated questionnaires will be completed and a subset of participants will participate in interviews. Study devices will be returned and participants will resume usual care.

Procedures for safety monitoring during trial:

Standard operating procedures for monitoring and reporting of all adverse events and adverse device events will be in place, including serious adverse events (SAE), serious adverse device effects (SADE) and specific adverse events (AE) such as severe hypoglycaemia.

A data monitoring and ethics committee (DMEC) will be informed of all serious adverse events and any unanticipated adverse device/method effects that occur during the study and will review compiled adverse event data at periodic intervals.

Criteria for withdrawal of subjects on safety grounds:

A participant may terminate participation in the study at any time without necessarily giving a reason and without any personal disadvantage.

The following pre-randomisation withdrawal criteria will apply:

* Participant time in range of >80% over the baseline masked CGM period
* Participant unable to demonstrate safe use of CGM as judged by the investigator

An investigator can stop the participation of a subject after consideration of the benefit/risk ratio. Possible pre- and post-randomisation withdrawal criteria include:

* Participant is unable to demonstrate safe use of study CGM and/or insulin pump as judged by the investigator
* Significant protocol violation or non-compliance
* Recurrent severe hypoglycaemia events related to use of the closed-loop system
* Recurrent severe persistent hyperglycaemia unrelated to infusion site failure and related to use of the closed-loop system
* Decision by the investigator or sponsor that termination is in the subject's best medical interest
* Allergic reaction to insulin
* Severe allergic reaction to adhesive surface of infusion set or glucose sensor
* Serious adverse events
* Pregnancy, planned pregnancy, or breast feeding
* Technical grounds (e.g. participant relocates)

ELIGIBILITY:
Inclusion Criteria:

1. Participant has cystic fibrosis related diabetes requiring insulin therapy for >3 months.
2. The participant is 16 years of age or older
3. Baseline time in target glucose range <80%
4. FEV1 >30% of predicted mean for age, sex, race, and height (equations of the Global Lung Function Initiative [GLI]) at the screening visit or within the past 6 months
5. Participant is willing to wear / carry study devices 24/7 (CGM / insulin pump / smartphone)
6. Participant is willing to follow study specific instructions

Exclusion Criteria:

1. Any physical or psychological disease or condition likely to interfere with the normal conduct of the study or interpretation of study results as judged by the investigator
2. Commencement of CFTR modulator therapy within previous 1 month
3. Previous solid organ transplant within the last 12 months or active on transplant waiting list
4. Use of closed-loop insulin therapy within the past 30 days
5. Known or suspected allergy to insulin
6. Severe visual impairment
7. Severe hearing impairment
8. Medically documented allergy or unable to tolerate the adhesive of plasters
9. Serious skin diseases at places of the body corresponding with sensor insertion sites
10. Participant is pregnant or breast feeding or planning pregnancy within next 12 months

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Time spent in the target glucose range between 3.9 and 10.0 mmol/L based on CGM glucose levels | 6 month intervention period

SECONDARY OUTCOMES:
Time spent with glucose >10.0 mmol/L based on CGM glucose levels | 6 month intervention period
  Key secondary endpoint
Mean glucose (mmol/L) based on CGM glucose levels | 6 month intervention period
  Key secondary endpoint
HbA1c | At 3 and 6 months
  Key secondary endpoint
Time spent with glucose levels <3.9 mmol/L based on CGM glucose levels | 6 month intervention period
Time spent with glucose levels <3.0 mmol/L based on CGM glucose levels | 6 month intervention period
Time spent with glucose levels <16.7 mmol/L based on CGM glucose levels | 6 month intervention period
Time in tighter glucose range 3.5 to 7.8 mmol/L based on CGM glucose levels | 6 month intervention period
Standard deviation of glucose based on CGM glucose levels | 6 month intervention period
Coefficient of variation of glucose based on CGM glucose levels | 6 month intervention period
Total daily insulin dose | 6 month intervention period
Total daily basal insulin dose | 6 month intervention period
Total daily bolus insulin dose | 6 month intervention period
Fasting C-peptide (pmol/L) | At 3 and 6 months
Body mass index (kg/m2) | At 3 and 6 months
Percentage of predicted FEV1 | At 3 and 6 months
Number of pulmonary exacerbations | 6 month intervention period
Number of hospitalisations | 6 month intervention period
Number of episodes of severe hypoglycaemia | 6 month intervention period
  Safety evaluation
Number of subjects experiencing severe hypoglycaemia | 6 month intervention period
  Safety evaluation
Frequency and nature of other adverse events or serious adverse events | 6 month intervention period
  Safety evaluation
Percentage of time of closed-loop operation | 6 month intervention period
  Utility evaluation
Percentage of time of CGM availability | 6 month intervention period
  Utility evaluation

OTHER OUTCOMES:
Human Factors Evaluation - Questionnaires | At 3 and 6 months
  Descriptive tabulations of questionnaires will be carried out, and scores will be calculated using provided scaling and scoring tools as appropriate.

CONTACTS AND LOCATIONS:
Locations (14):
- United Kingdom (14):
  - Belfast City Hospital, Belfast
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Royal Papworth Hospital, Cambridge
  - All Wales Adult CF Centre, Cardiff
  - Queen Elizabeth University Hospital, Glasgow
  - Glenfield Hospital, Leicester
  - Kings College Hospital, London
  - Royal Brompton Hospital, London
  - St Bartholomew's Hospital, London
  - Wythenshawe Hospital, Manchester University NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Southampton General Hospital, Southampton
  - Royal Stoke University Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication. To gain access, data requestors will need to sign a data access agreement.
  Fully anonymised data may be shared with third parties (EU or non-EU based) for the purposes of advancing management and treatment of diabetes.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to cb2000@medschl.cam.ac.uk and may be submitted up to 36 months following article publication.
Access Criteria: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to cb2000@medschl.cam.ac.uk and may be submitted up to 36 months following article publication.